CLINICAL TRIAL: NCT05155007
Title: A Phase 1, Open-label Study in Healthy Adult Participants to Assess the Effects of Ciclosporin Administration on the Single-dose Pharmacokinetics of Rilematovir
Brief Title: A Study in Healthy Adult Participants to Assess the Effects of Ciclosporin Administration on Rilematovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR109103; 2021-003801-23 (EudraCT Number); 53718678RSV1014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-12-08; First posted 2021-12-13 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-53718678; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will receive a single oral dose of rilematovir (Treatment A) in Treatment Period 1, followed by a single oral dose of ciclosporin (Treatment B) in Treatment Period 2 and then single oral dose of ciclosporin plus single oral dose of rilematovir (Treatment C) in Treatment Period 3 on Day 1 of each Treatment Period under fasted conditions. Each treatment period will be separated by a washout period of at least 5 days and maximum 21 days between subsequent intakes of study intervention.
  Interventions: Drug: Rilematovir; Drug: Ciclosporin
- Treatment Sequence BCA (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment C in Treatment Period 2 and then Treatment A in Treatment Period 3 on Day 1 of each Treatment Period under fasted conditions. Each treatment period will be separated by a washout period of at least 5 days and maximum 21 days between subsequent intakes of study intervention.
  Interventions: Drug: Rilematovir; Drug: Ciclosporin
- Treatment Sequence CAB (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment A in Treatment Period 2 and then Treatment B in Treatment Period 3 on Day 1 of each Treatment Period under fasted conditions. Each treatment period will be separated by a washout period of at least 5 days and maximum 21 days between subsequent intakes of study intervention.
  Interventions: Drug: Rilematovir; Drug: Ciclosporin
- Treatment Sequence ACB (Experimental): Participants will receive Treatment A in Treatment Period 1, followed by Treatment C in Treatment Period 2 and then Treatment B in Treatment Period 3 on Day 1 of each Treatment Period under fasted conditions. Each treatment period will be separated by a washout period of at least 5 days and maximum 21 days between subsequent intakes of study intervention.
  Interventions: Drug: Rilematovir; Drug: Ciclosporin
- Treatment Sequence BAC (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment A in Treatment Period 2 and then Treatment C in Treatment Period 3 on Day 1 of each Treatment Period under fasted conditions. Each treatment period will be separated by a washout period of at least 5 days and maximum 21 days between subsequent intakes of study intervention.
  Interventions: Drug: Rilematovir; Drug: Ciclosporin
- Treatment Sequence CBA (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment B in Treatment Period 2 and then Treatment A in Treatment Period 3 on Day 1 of each Treatment Period under fasted conditions. Each treatment period will be separated by a washout period of at least 5 days and maximum 21 days between subsequent intakes of study intervention.
  Interventions: Drug: Rilematovir; Drug: Ciclosporin

INTERVENTIONS:
Drug: Rilematovir — Rilematovir will be administered orally as per assigned treatment sequence.
  Other Names: JNJ-53718678
Drug: Ciclosporin — Ciclosporin will be administered orally as per assigned treatment sequence.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) of a single-dose of rilematovir co-administered with a single-dose of ciclosporin compared to a single-dose administration of rilematovir alone.

ELIGIBILITY:
Inclusion Criteria:

* Body weight not less than 50 kilograms (kg) and body mass index (BMI; weight kg/height^2 [meter {m^2}]) within the range 18.0 to 30.0 kilograms per meter square (kg/m^2) (inclusive)
* Female participants, except those that are of non-childbearing potential, must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test on Day -1 of Treatment Period 1
* A female participant using hormonal contraceptives as a means of birth control (a stable treatment for at least 30 days prior to screening) must agree to continue use of the same hormonal contraceptives throughout the study and for 90 days after the end of last study treatment
* Blood pressure (after the participant is supine for at least 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function, including: normal sinus rhythm (heart rate between 45 and 90 beats per minute, extremes included); QTc interval less than or equal to (<=) 450 milliseconds (ms) for men, <= 470 for women; QRS interval of less than (<) 110 ms; PR interval <= 200 ms; electrocardiogram morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* Participants with abnormal values for alanine aminotransferase (ALT) and aspartate aminotransferase (AST) Grade 1 or greater (greater than [>] 1.25* upper limit of normal [ULN])
* Participants with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Known allergies, hypersensitivity, or intolerance to rilematovir or its excipients. Known allergies, hypersensitivity, or intolerance to ciclosporin or its excipients
* Participant has received an experimental drug, vaccine or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study intervention is scheduled
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Treatment A and Treatment C: Maximum Observed Plasma Analyte Concentration (Cmax) of Rilematovir | Pre-dose up to 24 hours
  Cmax is defined as maximum observed plasma analyte concentration of rilematovir.
Treatment A and Treatment C: The Actual Sampling Time to Reach the Maximum Observed Plasma Analyte Concentration (Tmax) of Rilematovir | Pre-dose up to 24 hours
  Tmax is defined as the actual sampling time to reach the maximum observed plasma analyte concentration of rilematovir.
Treatment A and Treatment C: Apparent Terminal Elimination Half-life (T1/2) of Rilematovir | Pre-dose up to 96 hours
  T1/2 is defined as the apparent terminal elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve.
Treatment A and Treatment C: Area Under the Plasma Analyte Concentration Versus Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC[0-last]) of Rilematovir | Pre-dose up to 96 hours
  AUC(0-last) is defined as area under the plasma analyte concentration versus time curve from time zero to the time of the last measurable concentration of rilematovir.
Treatment A and Treatment C: Area Under the Plasma Analyte Concentration Versus Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Rilematovir | Pre-dose up to 96 hours
  AUC(0-infinity) is defined as area under the plasma analyte concentration versus time curve from time zero to infinite time of rilematovir.
Treatment A and Treatment C: Total Apparent Oral Clearance (CL/F) of Rilematovir | Pre-dose up to 96 hours
  CL/F is defined as total apparent oral clearance of rilematovir.

SECONDARY OUTCOMES:
Treatment B and Treatment C: Maximum Observed Whole Blood Analyte Concentration (Cmax) of Ciclosporin | Pre-dose up to 24 hours
  Cmax is defined as maximum observed whole blood analyte concentration of ciclosporin.
Treatment B and Treatment C: The Actual Sampling Time to Reach the Maximum Observed Whole Blood Analyte Concentration (Tmax) of Ciclosporin | Pre-dose up to 24 hours
  Tmax is defined as the actual sampling time to reach the maximum observed whole blood analyte concentration of ciclosporin.
Treatment B and Treatment C: Apparent Terminal Elimination Half-life (T1/2) of Ciclosporin | Pre-dose up to 96 hours
  T1/2 is defined as apparent terminal elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve.
Treatment B and Treatment C: Area Under the Whole Blood Analyte Concentration Versus Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC[0-last]) of Ciclosporin | Pre-dose up to 96 hours
  AUC(0-last) is defined as area under the whole blood analyte concentration versus time curve from time zero to the time of the last measurable concentration of ciclosporin.
Treatment B and Treatment C: Area Under the Whole Blood Analyte Concentration Versus Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Ciclosporin | Pre-dose up to 96 hours
  AUC(0-infinity) is defined as area under the whole blood analyte concentration versus time curve from time Zero to infinite time of ciclosporin.
Treatment B and Treatment C: Total Apparent Oral Clearance (CL/F) of Ciclosporin | Pre-dose up to 96 hours
  CL/F is defined as total apparent oral clearance of ciclosporin.
Percentage of Participants with Adverse Events (AEs) | Up to Week 12
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Percentage of Participants with Abnormalities in Electrocardiogram (ECG) | Up to Week 12
  Percentage of participants with abnormalities in ECG will be reported.
Percentage of Participants with Abnormalities in Physical Examination | Up to Week 12
  Percentage of participants with abnormalities in physical examination (including height, body weight and examination of all body systems and dermatologic examinations) will be reported.
Percentage of Participants with Abnormalities in Vital Signs | Up to Week 12
  Percentage of participants with abnormalities in vital signs (including temperature [tympanic], pulse/heart rate, blood pressure [systolic and diastolic]) will be reported.
Percentage of Participants with Abnormalities in Clinical Laboratory Tests | Up to Week 12
  Percentage of participants with abnormalities in clinical laboratory tests (including serum chemistry, hematology and routine urinalysis) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency